CLINICAL TRIAL: NCT06739278
Title: Analysis for the Efficacy of Individual Treatment of Perianal Fistulizing Crohn's Disease With Ustekinumab
Brief Title: Individual Treatment of Ustekinumab in Perianal Fistulizing Crohn's Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: SAHoWMU-CR2024-01-222
Record Dates: First submitted 2024-12-09; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study intends to further explore the actual efficacy of ustekinumab in the individualized treatment of anal fistula Crohn's disease.

DETAILED DESCRIPTION:
Participants in the study receive ustekinumab injections as part of routine medical care. The study just observes the efficacy retrospectively and does not interfere with treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Perianal Fistulizing Crohn's Disease
* Receive ustekinumab therapy

Exclusion Criteria:

* Ustekinumab combined with hormones, immunosuppressants, other biologics or small molecule drugs
* Combined with other autoimmune diseases, such as systemic lupus erythematosus, rheumatoid arthritis, Graves disease, etc.
* Combined with serious infectious diseases, such as active tuberculosis, EBV infection, cytomegalovirus infection, etc.
* Combined with malignant tumor
* Clinical data missing ≥30% or no follow-up

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with perianal fistulizing Crohn's disease
Sampling Method: Non-Probability Sample
Enrollment: 119 (Estimated)
Dates: Start 2024-12-20 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
imaging remission rate of anal fistula | Treatment week 0 to 32

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China